CLINICAL TRIAL: NCT01201863
Title: Neuroendocrine Dysfunction in Traumatic Brain Injury: Effects of Testosterone Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Cynthia Harrison-Felix, PhD, Director of Research, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10 IHA 11650
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Endocrine Dysfunction; Trauma; Brain Injury
Keywords: Testosterone; Traumatic Brain Injury; Hypogonadism; Endocrine Dysfunction; Low Testosterone in men with new Traumatic Brain Injury
MeSH Terms: conditions — Wounds and Injuries; Brain Injuries; Brain Injuries, Traumatic; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low T Intervention - Androgel Treatment (Experimental): Men with TBI meeting study criteria with Low Testosterone levels were randomly assigned to the Androgel treatment group. They underwent hormonal assays, FIM ratings and NIH Toolbox testing at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization.
  Interventions: Drug: Androgel (Testosterone Gel)
- Low T Intervention - Placebo Treatment (Placebo Comparator): Men with TBI meeting study criteria with Low Testosterone levels were randomly assigned to the Placebo gel treatment group. They underwent hormonal assays, FIM ratings and NIH Toolbox testing at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization.
  Interventions: Other: Placebo gel
- Normal T (No Intervention): A subset of men with TBI meeting study criteria with normal T at screening were assessed at all data collection time points to provide a control group. Thirty-eight men obtained normal T levels at screening of which 24 were followed.

INTERVENTIONS:
Drug: Androgel (Testosterone Gel) — 2.5 gram stickpacks administered with starting dosage of 5g increasing to a max of 10g.
  Arms: Low T Intervention - Androgel Treatment
Other: Placebo gel — 2.5 gram stickpacks with starting dose of 5g increasing to max of 10g.
  Arms: Low T Intervention - Placebo Treatment

SUMMARY:
The purpose of this study was to address 3 short term objectives; (1) Determine the effects of physiologic testosterone (T) therapy on neurological function and functional independence following traumatic brain injury (TBI) in hypogonadal men during inpatient rehabilitation; (2) Document the natural history of neuroendocrine dysfunction and recovery in men during inpatient rehabilitation after TBI; (3) Obtain data to validate the NIH toolbox, a novel assessment of neurological function for use in the TBI population; and 2 long-term objectives: (1) Utilize study findings to design a multicenter trial to further assess the impact of T therapy in hypogonadal men following TBI and (2) Impact TBI practice management with new information about neuroendocrine dysfunction after TBI and hormone treatments to improve outcomes.

DETAILED DESCRIPTION:
This randomized, double blind, placebo-controlled pilot study assessed the hormonal status of men on admission to an inpatient TBI rehabilitation program. 498 consecutively admitted men for TBI rehabilitation were screened for participation in the study. 22 participants with low T who met all criteria were randomized into placebo (n=10), or physiologic T therapy (n=12). Of those with normal T who met all criteria, 24 were randomized into a follow up group. All participants were evaluated every two weeks for up to 12 weeks: hormone levels, FIM ratings and NIH Toolbox testing as able. There was participant drop out over time as participants were discharged from the hospital. The final analysis examined differences between the normal T, low T Treatment and low T placebo groups on hormone levels, FIM ratings and NIH Toolbox results at baseline and weeks 2, 4 and 6.

ELIGIBILITY:
Inclusion Criteria:

1. History of TBI as defined as "damage to brain tissue caused by an external mechanical force as evidenced by loss of consciousness or post traumatic amnesia (PTA) due to brain trauma or by objective neurological findings that can be reasonably attributed to TBI on physical examination or mental status examination;"82
2. Moderate to severe TBI as indicated by a Glasgow Coma Scale (GCS) score of less than or equal to 12 at emergency department admission, or post traumatic amnesia (PTA) of greater than or equal to seven days post-injury, or radiographic evidence of intracranial injury;
3. Continuously hospitalized from time of injury until admission for rehabilitation;
4. Enrolled in study within 6 months of TBI;
5. Receiving inpatient rehabilitation for TBI at Craig Hospital;
6. Males between the ages of 16 to 65 (inclusive);
7. Approval by attending physician;
8. Testosterone level below the assay normal range;
9. Consent to study participation

   Exclusion Criteria:
10. History of any conditions that would prohibit testing contained in the NIH toolbox;
11. Non-English or non-Spanish speaking (to the extent that would limit the ability to complete study measures);
12. History of prior psychiatric illness requiring hospitalization;
13. Prior testosterone therapy;
14. History of or current or suspected hormonally dependent cancer , including carcinoma of the breast or prostate cancer;
15. Known hypersensitivity to any T gel ingredients including alcohol and soy products;
16. Hematocrit (HCT) greater than 55% (normal range in Colorado is up to 52) or transaminase elevation >4x upper limit of the normal range.
17. Abnormal finding on digital rectal examination such as nodule, asymmetry, or induration (Does not include enlarged prostate or abnormal rectal tone)
18. PSA>4.0
19. BMI <16 or >40kg/m2
20. History of untreated prolactinoma
21. History of severe heart failure or uncontrolled medical problem that would interfere with the participant's safety in the study as determined by the investigator.

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ripley, MD, Principal Investigator — Rehab Institute of Chicago
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

REFERENCES:
- [Result] Ripley DL, Gerber D, Pretz C, Weintraub AH, Wierman ME. Testosterone replacement in hypogonadal men during inpatient rehabilitation following traumatic brain injury: Results from a double-blind, placebo-controlled clinical pilot study. NeuroRehabilitation. 2020;46(3):355-368. doi: 10.3233/NRE-192992. PMID 32250330
- See also: Pubmed link to Testosterone replacement in hypogonadal men during inpatient rehabilitation following traumatic brain injury — http://pubmed.ncbi.nlm.nih.gov/32250330/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male in-patients with TBI at Craig Hospital meeting study criteria were screened from November 1, 2010 through July 24, 2014:
Pre-assignment Details: A total of 46 participants meeting all criteria were enrolled and randomized of which 22 had low testosterone levels, and 24 who had normal T were followed as controls. The total number who started and were followed was 46.
Groups:
- Intervention - Treatment: Men with TBI meeting study criteria with Low Testosterone levels will be randomly assigned to either a treatment or placebo group. They will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure.
  Androgel (Testosterone Gel): 2.5 gram stickpacks administered with starting dosage of 5g increasing to a max of 10g.
- Intervention Placebo: Men with TBI meeting study criteria with Low Testosterone levels will be randomly assigned to either a treatment or placebo group. They will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure.
  Androgel Placebo: 2.5 gram stickpacks with starting dose of 5g increasing to max of 10g.
- Normal - No Intervention: Enrolled participants with normal T
Period: Overall Study
Arm/Group | Intervention - Treatment | Intervention Placebo | Normal - No Intervention
Started | 12 | 10 | 24
Completed | 11 | 6 | 18
Not Completed | 1 | 4 | 6

BASELINE CHARACTERISTICS:
Population: 1 administrative withdrawal in Normal T Followed group making the total followed 46.
Groups:
- Low T Intervention - Treatment: Men with TBI meeting study criteria with Low Testosterone levels were randomly assigned to either a treatment or placebo group. They will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure.
  Androgel (Testosterone Gel): 2.5 gram stickpacks administered with starting dosage of 5g increasing to a max of 10g.
- Low T Intervention - Placebo: Men with TBI meeting study criteria with Low Testosterone levels were randomly assigned to either a treatment or placebo group. They will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure.
  Androgel Placebo: 2.5 gram stickpacks with starting dose of 5g increasing to max of 10g.
- Normal T No Intervention - Followed: A subset of men with TBI meeting study criteria with Normal Testosterone levels were assessed at all data collection time points. They will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure.
- Total: Total of all reporting groups
Arm/Group | Low T Intervention - Treatment | Low T Intervention - Placebo | Normal T No Intervention - Followed | Total
Number analyzed (Participants) | 12 | 10 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 24 | 46
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 12 | 10 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Restricted Functional Independence Measure (FIM)
Description: The FIM is the most widely accepted functional assessment measure in use in the rehabilitation community in the US. It is an 18-item ordinal clinician rating scale that is useful for assessment of functional skills progress during inpatient rehabilitation. It measures levels of independent/dependent performance of 13 motor functions and 5 cognitive functions. By adding the points for each item, the possible total score ranges from 18 to 126, with higher numbers indicating better performance. A restricted FIM total score that eliminated the toileting, bladder management and bowel management items was computed and used in the final analysis with scores ranging from 14-105). The restricted FIM total score was used as the primary outcome measure.
Time Frame: Administered at baseline and every other week for up to 12 weeks with 7 total possible administrations.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Intervention - Treatment: Men with TBI meeting study criteria with Low Testosterone levels were randomly assigned to either a treatment or placebo group. They participated in blood assays at baseline and every other week for up to 12 weeks during inpatient rehabilitation hospitalization. At the same assessment points, they were also scored on the FIM (primary outcome measure) and were administered the NIH Toolbox (Secondary Outcome Measure).
  Androgel (Testosterone Gel): 2.5 gram stickpacks administered with starting dosage of 5g increasing to a max of 10g.
- Intervention Placebo: Men with TBI meeting study criteria with Low Testosterone levels were randomly assigned to either a treatment or placebo group. They participated in blood assays at baseline and every other week for up to 12 weeks during inpatient rehabilitation hospitalization. At the same assessment points, they were also scored on the FIM (primary outcome measure) and were administered the NIH Toolbox (Secondary Outcome Measure).
  Androgel Placebo: 2.5 gram stickpacks with starting dose of 5g increasing to max of 10g.
- No Intervention: Men with TBI and normal T were followed for assessments only. They participated in blood assays at baseline and every other week for up to 12 weeks during inpatient rehabilitation hospitalization. At the same assessment points, they were also scored on the FIM (primary outcome measure) and were administered the NIH Toolbox (Secondary Outcome Measure).
Arm/Group | Intervention - Treatment | Intervention Placebo | No Intervention
Number analyzed (Participants) | 11 | 6 | 18
units on a scale
  Baseline | 34 [14 to 61] | 16 [14 to 29] | 21 [14 to 59]
  Six Week | 52 [22 to 98] | 31 [20 to 73] | 36 [14 to 94]
Statistical Analysis 1: Comparison: Intervention - Treatment vs Intervention Placebo; To investigate a difference in change in outcome over time between treatment and control, a trend analysis was used in place of a profile analysis, where both control and treatment arms are described more parsimoniously i.e. by a slope (change in outcome over time) (Fitzmaurice 2011); Test type: Superiority or Other; p = 0.9540, comparison of slopes; Slopes by group and slope difference; Slope = 0.07816, Standard Error of Mean 1.3315

ADVERSE EVENTS:
Groups:
- Low T Intervention - Treatment: Men with TBI meeting study criteria with Low Testosterone levels will be randomly assigned to either a treatment or placebo group. They will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure).
  Androgel (Testosterone Gel): 2.5 gram stickpacks administered with starting dosage of 5g increasing to a max of 10g.
- Low T Intervention - Placebo: Men with TBI meeting study criteria with Low Testosterone levels will be randomly assigned to either a treatment or placebo group. They will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure).
  Androgel Placebo: 2.5 gram stickpacks with starting dose of 5g increasing to max of 10g.
- Normal T - No Intervention: A subset of men with TBI meeting study criteria with Normal Testosterone levels will participate in blood assays at baseline and every other week for 12 weeks during inpatient rehabilitation hospitalization. They will also be scored on the FIM (primary outcome measure) and the NIH Toolbox (Secondary Outcome Measure).
Arm/Group | Low T Intervention - Treatment | Low T Intervention - Placebo | Normal T - No Intervention
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/24
Other Adverse Events (participants affected / at risk) | 2/13 | 3/10 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low T Intervention - Treatment (N=13) | Low T Intervention - Placebo (N=10) | Normal T - No Intervention (N=24)
Elevated ALT (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
greater than 100 ng/dl total testosterone change from screen to baseline (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0)
Elevated PSA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No